CLINICAL TRIAL: NCT05600894
Title: Venetoclax In Combination With ASTX727, an All-ORal TherapY for Chronic Myelomonocytic Leukemia and Other MDS/MPN With Excess Blasts (VICTORY-MDS/MPN): a Randomized, Phase 2 Trial
Brief Title: Venetoclax in Combination With ASTX727 for the Treatment of Chronic Myelomonocytic Leukemia and Other Myelodysplastic Syndrome/Myeloproliferative Neoplasm
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-08797; NCI-2022-08797 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10538 (Other: Yale University Cancer Center LAO); 10538 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts; Myelodysplastic/Myeloproliferative Neoplasm; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders | interventions — Specimen Handling; Biopsy; decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ASTX727, venetoclax) (Experimental): Patients receive ASTX727 PO QD on days 1-5 of each cycle and venetoclax PO QD on days 1-14 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy and aspiration and collection of blood samples throughout the study and undergo buccal swab sample collection at screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- Arm II (ASTX727) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not have response to treatment may cross over to Arm I. Patients also undergo bone marrow biopsy and aspiration and collection of blood samples throughout the study and undergo buccal swab sample collection at screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and buccal samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm I (ASTX727, venetoclax)

SUMMARY:
This phase II trial tests whether decitabine and cedazuridine (ASTX727) in combination with venetoclax work better than ASTX727 alone at decreasing symptoms of bone marrow cancer in patients with chronic myelomonocytic leukemia (CMML), myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) with excess blasts. Blasts are immature blood cells. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. The combination of ASTX727 and venetoclax may be more effective in reducing the cancer signs and symptoms in patients with CMML, or MDS/MPN with excess blasts.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the complete remission rates of ASTX727 and ASTX727 plus venetoclax in subjects with CMML and non-CMML MDS/MPN with excess (>= 5%) blasts.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (complete response [CR] + partial response [PR] + marrow response with erythroid response) of ASTX727 versus ASTX727 + venetoclax in this patient population.

II. To determine the overall survival, progression-free survival, allogeneic hematopoietic stem cell transplantation rate, clearance of the malignant clone, clonality at time of hematologic remission, number of red cell and platelet transfusions required and toxicity of ASTX727 versus ASTX727 + venetoclax.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (COMBINATION THERAPY): Patients receive ASTX727 orally (PO) once daily (QD) on days 1-5 of each cycle and venetoclax PO QD on days 1-14 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy and aspiration and collection of blood samples throughout the study and undergo buccal swab sample collection at screening.

ARM II (MONO THERAPY): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not have response to treatment may cross over to Arm I. Patients also undergo bone marrow biopsy and aspiration and collection of blood samples throughout the study and undergo buccal swab sample collection at screening.

After completion of study treatment, patients are followed up every 6 months for 5 years or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of an MDS/MPN "overlap" syndrome with >= 5% marrow blasts (including monocytic blast equivalent in case of CMML). Hydroxyurea may be used to control counts up until the start of therapy
* White blood cell (WBC) < 25,000/mm^3. Treatment with hydroxyurea is permitted to lower the WBC to reach this criterion
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ASTX727 in combination with venetoclax in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless considered due to Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN OR =< 5.0 x institutional ULN for patients with liver metastases
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Hormonal therapy for prior or concurrent malignancy is allowed
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) and/or family member available will also be eligible
* Ability to swallow pills

Exclusion Criteria:

* Patients with need for emergent disease-directed therapy excluding hydroxyurea
* More than one cycle of previous MDS/MPN-directed therapy, or MDS-directed therapy including lenalidomide and hypomethylating agent (HMAs) such as decitabine or azacitidine, excluding hydroxyurea. Prior use of erythropoietin stimulating agents (ESA) and thrombopoietic agents is allowed, but must be discontinued 4 weeks prior to study treatment
* Patients currently or previously receiving an investigational agent or device within 4 weeks of the first dose of treatment
* Patients with symptomatic uncontrolled central nervous system (CNS) disease. Imaging to confirm the absence of brain metastases is not required. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Patients who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit within 3 days prior to the initiation of study treatment and are unwilling to discontinue consumption of these throughout the receipt of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ASTX727 or venetoclax
* Patients with uncontrolled intercurrent illness (e.g. requiring intravenous therapy) at the discretion of the investigator
* Pregnant women are excluded from this study because venetoclax and ASTX727 have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, breastfeeding should be discontinued if the mother is treated with venetoclax. These potential risks may also apply to other agents used in this study. Patients must be post-menopausal or with evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1

  * Post-menopausal is defined as:

    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50 years of age
    * Radiation-induced oophorectomy with last menses > 1 year ago
    * Chemotherapy-induced menopause with > 1 year interval since last menses
    * Surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women of child-bearing potential must agree to use adequate contraception (hormonal birth control or abstinence) prior to study entry and for the duration of study participation, and for 6 months following completion of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception (latex or synthetic condom or abstinence) prior to the study, for the duration of study participation, and 3 months after completion of venetoclax and ASTX727 administration
* Patients with any other medical condition for which the expected survival is below 12 months
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or assessment of the investigational regimen
* Patients with uncontrolled infection at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Up to 4 cycles
  The complete remission rate will be compared between two arms using Fisher's exact test. Logistical regression will be used to estimate the effect of combination treatment on complete remission adjusting for covariates of interest.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization until death from any cause, assessed up to 5 years
  Will be calculated using the Kaplan-Meier method. Comparisons of OS between treatment arms will be conducted using the one-sided log-rank test. Hazard ratios will be computed using the Cox proportional hazards model. The censored follow-up time for patients without death information is the date of last contact.
Progression-free survival (PFS) | From randomization until disease progression or death from any cause, whichever comes first, assessed up to 5 years
  Will be calculated using the Kaplan-Meier method. Comparisons of PFS between treatment arms will be conducted using the one-sided log-rank test. Hazard ratios will be computed using the Cox proportional hazards model. For patients alive without progression, PFS will be censored at the date of the last disease evaluation.
Incidence of adverse events | Up to 5 years
  An undesired effect of a drug or other type of treatment, such as surgery. Adverse events can range from mild to severe and can be life-threatening.

CONTACTS AND LOCATIONS:
Overall Officials: Rory M Shallis, Principal Investigator — Yale University Cancer Center LAO
Locations (34):
- United States (33):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UCI Health Laguna Hills, Laguna Hills, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm